CLINICAL TRIAL: NCT02804672
Title: Study on Cardiovascular Health, Nutrition and Frailty in Older Adults in Spain
Acronym: Seniors-ENRICA
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Fernando Rodríguez-Artalejo, Professor of Preventive Medicine and Public Health, Universidad Autonoma de Madrid
Other Study IDs: Seniors-ENRICA
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Physical Disability; Cardiovascular Risk Factors
Keywords: Cardiovascular health; Diet; Functional limitations; Frailty; Older adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examine the association between ideal cardiovascular health, diet and other lifestyles, biological risk factors, either well-established or emergent, and the risk of frailty in older adults, throughout different waves (2008-10, 2012 and 2015 -16).

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized Spanish resident
* 60 years and over

Exclusion Criteria:

* None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-living individuals in Spain aged 60 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 1566 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Frailty | 3 years
  Method of assessment: Fried criteria

SECONDARY OUTCOMES:
Change from baseline in Cardiovascular health | 3 years
  Method of assessment: 7 cardiovascular health metrics as defined by American Heart Association

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rodríguez-Artalejo, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health, Universidad Autónoma de Madrid; Jose R Banegas, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health, Universidad Autónoma de Madrid
Locations (1):
- Department of Preventive Medicine and Public Health, Universidad Autónoma de Madrid, Madrid, Spain

REFERENCES:
- [Result] Banegas JR, de la Cruz JJ, Graciani A, Lopez-Garcia E, Gijon-Conde T, Ruilope LM, Rodriguez-Artalejo F. Impact of Ambulatory Blood Pressure Monitoring on Reclassification of Hypertension Prevalence and Control in Older People in Spain. J Clin Hypertens (Greenwich). 2015 Jun;17(6):453-61. doi: 10.1111/jch.12525. Epub 2015 Mar 16. PMID 25779903
- [Result] Garcia-Esquinas E, Graciani A, Guallar-Castillon P, Lopez-Garcia E, Rodriguez-Manas L, Rodriguez-Artalejo F. Diabetes and risk of frailty and its potential mechanisms: a prospective cohort study of older adults. J Am Med Dir Assoc. 2015 Sep 1;16(9):748-54. doi: 10.1016/j.jamda.2015.04.008. Epub 2015 May 16. PMID 25986874
- [Result] Lana A, Rodriguez-Artalejo F, Lopez-Garcia E. Dairy Consumption and Risk of Frailty in Older Adults: A Prospective Cohort Study. J Am Geriatr Soc. 2015 Sep;63(9):1852-60. doi: 10.1111/jgs.13626. Epub 2015 Aug 27. PMID 26311353
- [Result] Sandoval-Insausti H, Perez-Tasigchana RF, Lopez-Garcia E, Garcia-Esquinas E, Rodriguez-Artalejo F, Guallar-Castillon P. Macronutrients Intake and Incident Frailty in Older Adults: A Prospective Cohort Study. J Gerontol A Biol Sci Med Sci. 2016 Oct;71(10):1329-34. doi: 10.1093/gerona/glw033. Epub 2016 Mar 4. PMID 26946103
- [Result] Graciani A, Garcia-Esquinas E, Lopez-Garcia E, Banegas JR, Rodriguez-Artalejo F. Ideal Cardiovascular Health and Risk of Frailty in Older Adults. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):239-45. doi: 10.1161/CIRCOUTCOMES.115.002294. Epub 2016 May 10. PMID 27166207
- [Derived] Vazquez-Fernandez A, Caballero FF, Yevenes-Briones H, Struijk EA, Baylin A, Fung TT, Lopez-Garcia E. Plant and Animal Protein Intake and Transitions From Multimorbidity to Frailty and Mortality in Older Adults. J Cachexia Sarcopenia Muscle. 2025 Feb;16(1):e13729. doi: 10.1002/jcsm.13729. PMID 39971333
- [Derived] Marcos-Delgado A, Yevenes-Briones H, Fernandez-Villa T, Martin-Sanchez V, Guallar-Castillon P, Rodriguez-Artalejo F, Lopez-Garcia E. Association between diet quality and malnutrition: pooled results from two population-based studies in older adults. BMC Geriatr. 2024 May 10;24(1):417. doi: 10.1186/s12877-024-04984-5. PMID 38730363
- [Derived] Delgado-Velandia M, Maroto-Rodriguez J, Ortola R, Garcia-Esquinas E, Rodriguez-Artalejo F, Sotos-Prieto M. Plant-Based Diets and All-cause and Cardiovascular Mortality in a Nationwide Cohort in Spain: The ENRICA Study. Mayo Clin Proc. 2022 Nov;97(11):2005-2015. doi: 10.1016/j.mayocp.2022.06.008. PMID 36333014
- [Derived] Sotos-Prieto M, Ortola R, Lopez-Garcia E, Rodriguez-Artalejo F, Garcia-Esquinas E. Adherence to the Mediterranean Diet and Physical Resilience in Older Adults: The Seniors-ENRICA Cohort. J Gerontol A Biol Sci Med Sci. 2021 Feb 25;76(3):505-512. doi: 10.1093/gerona/glaa277. PMID 33152061
- [Derived] Garcia-Esquinas E, Rodriguez-Sanchez I, Ortola R, Lopez-Garcia E, Caballero FF, Rodriguez-Manas L, Banegas JR, Rodriguez-Artalejo F. Gender Differences in Pain Risk in Old Age: Magnitude and Contributors. Mayo Clin Proc. 2019 Sep;94(9):1707-1717. doi: 10.1016/j.mayocp.2019.03.034. PMID 31486377
- [Derived] Sandoval-Insausti H, Blanco-Rojo R, Graciani A, Lopez-Garcia E, Moreno-Franco B, Laclaustra M, Donat-Vargas C, Ordovas JM, Rodriguez-Artalejo F, Guallar-Castillon P. Ultra-processed Food Consumption and Incident Frailty: A Prospective Cohort Study of Older Adults. J Gerontol A Biol Sci Med Sci. 2020 May 22;75(6):1126-1133. doi: 10.1093/gerona/glz140. PMID 31132092